CLINICAL TRIAL: NCT05231187
Title: T2Resistance 510(k) Study Protocol - Detection and Identification of Several Classes of Resistance Genes in Both Gram-positive and Gram-negative Pathogens
Brief Title: T2Resistance - Detection of Resistance Related Genes
Status: Completed | Type: Observational
Sponsor: T2 Biosystems (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 210-11147
Record Dates: First submitted 2022-01-28; First posted 2022-02-09 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Resistance Bacterial
Keywords: Antibiotic resistant markers

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood Samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Prospective Arm: Subjects has had a diagnostic blood culture ordered per routine standard of care.
  Interventions: Diagnostic Test: T2Resistance Panel
- Contrived Arm: Samples of healthy whole blood spiked with bacterial strains harboring the resistance gene targets on the T2Resistance Panel.
  Interventions: Diagnostic Test: T2Resistance Panel
- Healthy Donor Arm: Healthy donor subjects.
  Interventions: Diagnostic Test: T2Resistance Panel

INTERVENTIONS:
Diagnostic Test: T2Resistance Panel — The T2Resistance Panel is an in vitro diagnostic medical device that runs on the T2Dx instrument and detects bacterial markers that are commonly associated with antibiotic resistance. T2Resistance Panel detects thirteen (13) markers of resistance in seven detection channels:
  1. blaKPC
  2. blaCTX-M
  3. blaNDM / blaVIM / blaIMP
  4. blaOXA-48 Group
  5. vanA / vanB
  6. mecA / mecC
  7. AmpC (blaCMY / blaDHA)

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the T2Resistance Panel by validating clinical performance in three study arms:

1. Prospective arm: positive percent agreement (PPA) and negative percent agreement (NPA) against genetic determinants of resistance detected in whole blood clinical samples or isolates collected from positive blood cultures prospectively collected clinical samples of whole blood.
2. Contrived arm: positive percent agreement (PPA) and negative percent agreement (NPA) against samples with known status, via spiking healthy whole blood samples with bacterial strains harboring the resistance gene targets on the T2Resistance Panel.
3. Healthy donor arm: negative percent agreement (NPA) with presumed negativity of healthy donor whole blood samples.

The data from all arms of the study will be used to support the Premarket Notification for the T2Resistance Panel to the U.S. Food and Drug Administration.

Primary Endpoints

The primary endpoints of this study with the T2Resistance Panel are estimated sensitivity, specificity, and safety.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and effectiveness of the T2Resistance Panel by validating clinical performance in three study arms:

1. Prospective arm: positive percent agreement (PPA) and negative percent agreement (NPA) against genetic determinants of resistance detected in whole blood clinical samples or isolates collected from positive blood cultures prospectively collected clinical samples of whole blood.
2. Contrived arm: positive percent agreement (PPA) and negative percent agreement (NPA) against samples with known status, via spiking healthy whole blood samples with bacterial strains harboring the resistance gene targets on the T2Resistance Panel.
3. Healthy donor arm: negative percent agreement (NPA) with presumed negativity of healthy donor whole blood samples.

The data from all arms of the study will be used to support the Premarket Notification for the T2Resistance Panel to the U.S. Food and Drug Administration.

Primary Endpoints

The primary endpoints of this study with the T2Resistance Panel are estimated sensitivity, specificity, and safety.

Sensitivity

The estimated sensitivity of the T2Resistance Panel will be derived from two metrics:

1. Prospective arm: positive concordance between a positive result on the T2Resistance Panel and a positive sequencing result from a whole blood sample or isolate from positive blood culture
2. Contrived arm: positive concordance between a positive result on the T2Resistance Panel and a sample spiked with a bacterial isolates sequence confirmed to be harboring a known resistance gene on the T2Resistance Panel.

The Contrived arm of the study will consist of ≥ 350 whole blood samples spiked with titer levels ranging from < 1 CFU/mL to 100 CFU/mL. These samples will be provided to selected test sites for testing. Sensitivity values will be calculated separately for each channel and study arm, e.g., Prospective and Contrived study arms for blaKPC, blaCTX-M, blaNDM / blaVIM / blaIMP, blaOXA-48 Group, vanA / vanB, mecA / mecC and AmpC (blaCMY / blaDHA) channels.

Specificity

The estimated specificity of the T2Resistance Panel will be derived from three metrics:

1. Prospective arm: negative concordance between a negative ("Target not Detected") result on the T2Resistance Panel and a negative sequencing result from whole blood sample or isolate from positive blood culture
2. Healthy donor arm: negative concordance between a negative ("Target not Detected") result on the T2Resistance Panel and a presumed negativity of healthy donor whole blood sample
3. Contrived arm: negative concordance between a negative ("Target not Detected") result in a given channel of the T2Resistance Panel and the presence of a spiked bacteria known to not harbor the given resistance gene on the T2Resistance Panel

Specificity values will be calculated separately for each channel and study arm, e.g., Prospective, Healthy donor, and Contrived study arms for blaKPC, blaCTX-M, blaNDM / blaVIM / blaIMP, blaOXA-48 Group, vanA / vanB, mecA / mecC and AmpC (blaCMY / blaDHA) channels.

Safety

There are no expected adverse events that are directly related to the T2Resistance Panel and the T2Dx Instrument as a result of participating in this study. Since the device does not come in contact with the patients and the test results are not used in clinical practice as part of standard of care, the only adverse events associated with study participation is the collection of blood samples for T2Resistance Panel testing.

ELIGIBILITY:
Inclusion Criteria:

Prospective Arm:

* Obtain informed consent according to institutional requirements, as needed.
* Patient has had a diagnostic blood culture ordered per routine standard of care.
* Patient is 18 years of age or older.

Exclusion Criteria:

Prospective Arm

* Patient has other co-morbid condition(s) that, in the opinion of the Investigator, could limit the patient's ability to participate in the study or impact the scientific integrity of the study.
* Patient has had previous specimens tested for the T2Resistance Panel with valid results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting at the Investigational Site (Hospital, Clinical) and having a diagnostic blood culture ordered per routine standard of care.
Sampling Method: Probability Sample
Enrollment: 1566 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
Sensitivity - Prospective | Six months from collection, maximum.
  Positive concordance between positive T2Resistance panel results for positive samples.
Specificity - Prospective | Six months from collection, maximum.
  Negative concordance between a negative ("Target not Detected") result on the T2Resistance Panel and a negative sequencing result or a known negative sample.
Safety / Adverse Events | During patient blood draw or immediately after blood draw, typically <1 hour.
  Potential adverse events associated with the collection of blood samples for T2Resistance Panel Testing.

SECONDARY OUTCOMES:
Sensitivity - Contrived | Six months from collection, maximum.
  Concordance between T2Resistance Panel results and positive blood culture, and contrived samples.
Specificity - Contrived | Six months from collection, maximum.
  Concordance between a negative ("Target not Detected") result on the T2Resistance Panel and sensitivity results associated with antibiotic susceptibility testing from positive blood culture samples or positive contrived samples.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Smith, Ph.D., Study Director — T2 Biosystems
Locations (10):
- United States (10):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - Tampa General Hospital, Tampa, Florida
  - Ochsner Medical Center, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - University Health, Truman Medical Center, Kansas City, Missouri
  - New York University Langone Health, Brooklyn, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Texas Health Science Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No